CLINICAL TRIAL: NCT06265350
Title: Cryoablation Combined With Cardonilizumab and Bevacizumab in Hepatocellular Carcinoma With Pulmonary Metastases: A Single-center, Prospective, Randomized Controlled Phase II Study
Brief Title: Cryoablation Combined With Cardonilizumab and Bevacizumab in Hepatocellular Carcinoma With Pulmonary Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liver Project 5
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer Stage IV; Pulmonary Metastases; Cadonilimab; Bevacizumab; Cryoablation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Bevacizumab; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab+Cadonilimab group (Active Comparator): Patients accepted Bevacizumab (7.5mg/kg，Q3W， IV) plus Cadonilimab (375mg，Q3W， IV)
  Interventions: Drug: Cadonilimab; Drug: Bevacizumab
- Cryoablation+Bevacizumab+Cadonilimab (Experimental): Patients accepted Cryoablation of pulmanary metastases combined with Bevacizumab (7.5mg/kg，Q3W， IV) and Cadonilimab (375mg，Q3W， IV)
  Interventions: Drug: Cadonilimab; Drug: Bevacizumab; Procedure: Cryoablation

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab, 375mg，Q3W， IV
Drug: Bevacizumab — Bevacizumab, 7.5mg/kg，Q3W， IV
Procedure: Cryoablation — Patients accepted Cryoablation of pulmanary metastases
  Arms: Cryoablation+Bevacizumab+Cadonilimab

SUMMARY:
This study intends to evaluate the efficacy and safety of cryoablation combined with Cardonilizumab and Bevacizumab in hepatocellular carcinoma with pulmonary metastases.

DETAILED DESCRIPTION:
For advanced hepatocellular carcinoma (HCC), the lung is the most common metastatic organ, accounting for 30-50% of extrahepatic diseases. The standard therapy for advanced HCC with lung metastases according to the Barcelona Clinic Liver Cancer (BCLC) criteria is system therapy.

However, studies have proven that palliative ablation could improve the tumor controlling effect and the outcomes.

Cryoablation is a treatment method that involves freezing tumors at extremely low temperatures to destroy and eliminate them. This therapeutic approach can result in the death of tumor cells through necrosis and also stimulate immune targeting of tumor cells. These immune responses occur as a result of tumor cell death caused by the ablation procedure. In comparison to conventional cancer therapies, cryoablation has minimal adverse reactions and has the potential to promote a more extensive and effective release of self-generated antigens into the bloodstream.

Targeting vascular endothelial growth factor (VEGF) could reduce VEGF-mediated immunosuppression within the tumor. The IMbrave150 study of atezolizumab and bevacizumab versus sorafenib demonstrated response rates of 29.8% vs 12%, respectively, and median overall survival of 19.8 months in the combination arm versus 13.4 months in the sorafenib (P <0.001). Bevacizumab could enhance anti-PD-1 and anti-programmed death ligand 1 (PD-L1) efficacy by reversing VEGF-mediated immunosuppression and promoting T-cell infiltration in tumors (2).

Cadonilimab is a first-in-class bispecific, humanized IgG1 antibody targeting PD-1 and CTLA-4, which has the potential to boost immune surveillance in tumors. Preclinical studies have shown that its tetravalent design enhances its high binding activity in the tumor microenvironment. With no Fc binding, Cadonilimab could eliminate a series of functions mediated by the Fc receptor, which contribute to a poor safety profile in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. primary or recurrent HCC;
2. synchronous metastases (within one month after diagnosing of HCC) or asynchronous metastases (more than one month after diagnosis of HCC);
3. pulmonary-only metastases >5 and ≤10;
4. metastases diameter ≤ 5 cm;
5. intrahepatic tumors ≤5, and tumor burden ≤1/2 liver volume;
6. PVTT type Vp≤3;
7. patients underwent first-line system therapy failure, the first-line system included tyrosine kinase inhibitor (TKI), such as Sorafenib or Lenvatinib, with or without PD-1 or PDL1 inhibitor;
8. the intrahepatic tumors were effectively controlled and pulmonary metastases were no progression, and the controlled intrahepatic tumors were defined as partial or stable response according to modified Response Evaluation Criteria in Solid Tumors (mRECIST);
9. locoregional therapy (including TACE or HAIC) were also included;
10. Child-Pugh class A or B;
11. PS 0 or 1;
12. no history of other malignancies.

Exclusion Criteria:

1. under 18 years or over 75 years;
2. metastases >10
3. non-lung metastases;
4. incomplete clinical data;
5. metastases diameter > 5 cm;
6. intrahepatic tumors > 5, and tumor burden > 1/2 liver volume;
7. PVTT type Vp 4;
8. lost to follow-up within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as partial response and complete response.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of inclusion to the date of the first objectively documented tumor progression or death due to any cause.
Overall survival (OS) | 12 months
  OS is the length of time from the date of inclusion until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimei Hunag, MD, Study Director — Sun Yat-sen University; Jinhua Huang, MD, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China